CLINICAL TRIAL: NCT06609135
Title: Relationship Between Electrical Impedance Tomography (EIT) Measurements and Parameters of Respiratory Status in Very Preterm Infants: An Observational Cohort Study
Brief Title: Relationship Between EIT and Respiratory Status in Very Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lawrence Rhein (Other)
Collaborators: SenTec AG, Ringstrasse 39, CH-4106 Therwil (Unknown)
Responsible Party: Sponsor-Investigator, Lawrence Rhein, Chair, Department of Pediatrics, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00001180
Record Dates: First submitted 2024-06-24; First posted 2024-09-24 (Actual); Results first posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Chronic Lung Disease of Prematurity; Bronchopulmonary Dysplasia; Premature Lungs
Keywords: Electrical Impedance Tomography (EIT); Prematurity; Pulmonary Function Testing; Noninvasive ventilation; Continuous Positive Airway Pressure (CPAP); Transcutaneous CO2 monitor (TCOM)
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Electrical Impedance Tomography (EIT) and CO2 monitor (Experimental): Participating infants will have the EIT belt placed at a minimum of twice per week throughout the NICU stay. A respiratory therapist or physician will place the EIT belt at the end of a feed and remove it at the next feed. A transcutaneous CO2 monitor will be placed concurrently.
  Interventions: Device: Sentec LuMon Device (EIT system); Device: Sentec Digital Monitoring System (transcutaneous CO2 monitor)

INTERVENTIONS:
Device: Sentec LuMon Device (EIT system) — Sentec EIT belts will be placed on infants up to once daily from consent through NICU discharge.
Device: Sentec Digital Monitoring System (transcutaneous CO2 monitor) — Sentec transcutaneous CO2 monitors will be placed on infants concurrently with EIT belts.

SUMMARY:
Electrical Impedance Tomography (EIT) is a non-invasive imaging technique that can measure lung function in real time. This study will follow premature infants to see if EIT can help predict which infants will be successful in weaning off respiratory support by 32-33 weeks gestational age. If successful, EIT could be used to develop new guidelines for respiratory support in premature infants.

ELIGIBILITY:
Inclusion Criteria:

* Infants admitted to the University of Massachusetts Memorial Medical Center (UMMMC) Neonatal Intensive Care Unit (NICU)
* Born between 25+0- and 29+6-weeks of gestation

Exclusion Criteria:

* Infants with major congenital anomalies
* Infants with severe hemodynamic instability

Min Age: 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-11-04 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Rhein, MD, MPH, Principal Investigator — UMASS Chan Medical School
Locations (1):
- UMASS Memorial Medical Center, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The EIT and TCOM data, study methodology may be valuable for other clinical investigators and thus worth sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The plan is to share all IPD the underlie the results of a publication within 6 months of publication.
Access Criteria: Requests by other clinical investigators will be reviewed by with Lawrence Rhein or Mohammad Jaber and if deemed reasonable IPD to be shared.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment period lasted from November 2023 through August 2024. Recruitment occured in the UMASS Memorial Medical Center NICU. 40 very preterm infants were screened, 37 were eligible, 33 were approached, and 20 were successfully enrolled.
Period: Overall Study
Arm/Group | Electrical Impedance Tomography (EIT) and CO2 Monitor
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Electrical Impedance Tomography (EIT) and CO2 Monitor
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 0 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
Birth Gestational Age [Mean (Standard Deviation); unit: weeks] | 28.2 (1.5)
Birth Weight [Mean (Standard Deviation); unit: grams] | 1124 (280)
Vaginal Delivery [Count of Participants; unit: Participants] | 9
Betamethasone complete [Count of Participants; unit: Participants] | 14
Postnatal Diuretics [Count of Participants; unit: Participants] | 3
Postnatal Steroids [Count of Participants; unit: Participants] | 4
Chronic Lung Disease of Prematurity [Count of Participants; unit: Participants] | 6

OUTCOME MEASURES:

1. Primary Outcome: EIT Metric Global Inhomogeneity Index at 31 Weeks Post Menstrual Age in Those Successful in Discontinuation of Non-invasive Ventilation at 32 Weeks Post Menstrual Age.
Description: The primary outcome is to determine whether electrical impedance tomography metrics, specifically Global Inhomogeneity Index (GI) and Functional Lung Space, measured at 31 weeks post menstrual age are associated with successful discontinuation of non-invasive ventilation at 32 weeks post menstrual age. GI, a measure of ventilation inhomogeneity, ranges from 0 (completely homogeneous) to 1 (completely inhomogeneous). Lower GI values are interpreted as better.
Time Frame: 3-hour continuous measurement semi-weekly from 28+0/7 weeks or 7 days postnatally if older than 27+1/7 weeks birth gestational age to establish baseline. Comparative measurement obtained between 30+5/7 and 31+2/7 weeks postmenstrual age=up to 1-3 weeks.
Population: Data at 31 weeks was available for 3 of the 6 infants that weaned to room air at 32 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Electrical Impedance Tomography (EIT) and CO2 Monitor
Number analyzed (Participants) | 3
score on a scale | 0.54 (0.03)
Statistical Analysis 1: Comparison: Electrical Impedance Tomography (EIT) and CO2 Monitor; Statistical Analysis assessed correlation of GI values at 31 weeks between participants that were successful in discontinuation of non-invasive ventilation at 32 weeks postmenstrual age and those that were unsuccessful; Test type: Superiority; p = 0.045, t-test, 2 sided

2. Primary Outcome: EIT Metric Global Inhomogeneity Index at 31 Weeks Post Menstrual Age in Those Unsuccessful in Discontinuation of Non-invasive Ventilation at 32 Weeks Post Menstrual Age.
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Data at 31 weeks was available for 8 of 14 infants that did not wean to room air at 32 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Electrical Impedance Tomography (EIT) and CO2 Monitor
Number analyzed (Participants) | 8
score on a scale | 0.7 (0.13)
Statistical Analysis 1: Comparison: Electrical Impedance Tomography (EIT) and CO2 Monitor; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.045, t-test, 2 sided

3. Secondary Outcome: EIT Metric Global Inhomogeneity Index at 32 Weeks Post Menstrual Age in Those Successful in Discontinuation of Non-invasive Ventilation at 33 Weeks Post Menstrual Age.
Description: The first secondary outcome is to determine whether electrical impedance tomography metrics, specifically Global Inhomogeneity Index and Functional Lung Space, measured at 32 weeks post menstrual age are associated with successful discontinuation of non-invasive ventilation at 33 weeks post menstrual age. GI, a measure of ventilation inhomogeneity, ranges from 0 (completely homogeneous) to 1 (completely inhomogeneous). Lower GI values are interpreted as better.
Time Frame: 3-hour continuous measurement semi-weekly from 28+0/7 weeks or 7 days postnatally if older than 27+1/7 weeks birth gestational age to establish baseline. Comparative measurement obtained between 31+5/7 and 32+2/7 weeks postmenstrual age=up to 2-4 weeks.
Population: Data at 32 weeks was available for all 4 infants that weaned to room air at 33 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Electrical Impedance Tomography (EIT) and CO2 Monitor
Number analyzed (Participants) | 4
score on a scale | 0.62 (0.1)
Statistical Analysis 1: Comparison: Electrical Impedance Tomography (EIT) and CO2 Monitor; Statistical Analysis assessed correlation of GI values at 32 weeks between participants that were successful in discontinuation of non-invasive ventilation at 33 weeks postmenstrual age and those that were unsuccessful; Test type: Superiority; p = 0.49, t-test, 2 sided

4. Secondary Outcome: EIT Metric Global Inhomogeneity Index at 32 Weeks Post Menstrual Age in Those Unsuccessful in Discontinuation of Non-invasive Ventilation at 33 Weeks Post Menstrual Age.
Description: as for outcome 3
Time Frame: as for outcome 3
Population: Data at 32 weeks was available for 6 of 10 infants that did not wean to room air at 33 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Electrical Impedance Tomography (EIT) and CO2 Monitor
Number analyzed (Participants) | 6
score on a scale | 0.67 (0.12)
Statistical Analysis 1: Comparison: Electrical Impedance Tomography (EIT) and CO2 Monitor; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.49, t-test, 2 sided

5. Secondary Outcome: EIT Metric Global Inhomogeneity Index at 34 Weeks Post Menstrual Age in Those Successful in Discontinuation of Non-invasive Ventilation at 36 Weeks Post Menstrual Age.
Description: The second secondary outcome is to determine whether electrical impedance tomography metrics, specifically Global Inhomogeneity Index and Functional Lung Space, measured at 34 weeks post menstrual age are associated with successful discontinuation of non-invasive ventilation at 36 weeks post menstrual age. GI, a measure of ventilation inhomogeneity, ranges from 0 (completely homogeneous) to 1 (completely inhomogeneous). Lower GI values are interpreted as better.
Time Frame: 3-hour continuous measurement semi-weekly from 28+0/7 weeks or 7 days postnatally if older than 27+1/7 weeks birth gestational age to establish baseline. Comparative measurement obtained between 33+5/7 and 34+2/7 weeks postmenstrual age=up to 4-6 weeks.
Population: Data at 34 weeks was available for 3 of the 4 infants that weaned to room air by 36 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Electrical Impedance Tomography (EIT) and CO2 Monitor
Number analyzed (Participants) | 3
score on a scale | 0.55 (0.1)
Statistical Analysis 1: Comparison: Electrical Impedance Tomography (EIT) and CO2 Monitor; Statistical Analysis assessed correlation of GI values at 34 weeks between participants that were successful in discontinuation of non-invasive ventilation by 36 weeks postmenstrual age and those that were unsuccessful; Test type: Superiority; p = 0.56, t-test, 2 sided

6. Secondary Outcome: EIT Metric Global Inhomogeneity Index at 34 Weeks Post Menstrual Age in Those Unsuccessful in Discontinuation of Non-invasive Ventilation at 36 Weeks Post Menstrual Age.
Description: as for outcome 5
Time Frame: as for outcome 5
Population: Data at 34 weeks was available for 4 of the 6 infants that did not wean to room air by 36 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Electrical Impedance Tomography (EIT) and CO2 Monitor
Number analyzed (Participants) | 4
score on a scale | 0.59 (0.09)
Statistical Analysis 1: Comparison: Electrical Impedance Tomography (EIT) and CO2 Monitor; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.56, t-test, 2 sided

7. Primary Outcome: EIT Metric Functional Lung Space at 31 Weeks Post Menstrual Age in Those Successful in Discontinuation of Non-invasive Ventilation at 32 Weeks Post Menstrual Age.
Description: The primary outcome is to determine whether electrical impedance tomography metrics, specifically Global Inhomogeneity Index (GI) and Functional Lung Space, measured at 31 weeks post menstrual age are associated with successful discontinuation of non-invasive ventilation at 32 weeks post menstrual age.
Time Frame: as for outcome 1
Population: Data at 31 weeks was available for 3 of the 6 infants that weaned to room air at 32 weeks
Measure: Mean (Standard Deviation); unit: percentage of total lung space
Arm/Group | Electrical Impedance Tomography (EIT) and CO2 Monitor
Number analyzed (Participants) | 3
percentage of total lung space | 85 (2)
Statistical Analysis 1: Comparison: Electrical Impedance Tomography (EIT) and CO2 Monitor; Statistical Analysis assessed correlation of FLS values at 31 weeks between participants that were successful in discontinuation of non-invasive ventilation at 32 weeks postmenstrual age and those that were unsuccessful; Test type: Superiority; p = 0.09, t-test, 2 sided

8. Primary Outcome: EIT Metric Functional Lung Space at 31 Weeks Post Menstrual Age in Those Unsuccessful in Discontinuation of Non-invasive Ventilation at 32 Weeks Post Menstrual Age.
Description: as for outcome 7
Time Frame: as for outcome 1
Population: Data at 31 weeks was available for 8 of the 14 infants that did not wean to room air at 32 weeks
Measure: Mean (Standard Deviation); unit: percentage of total lung space
Arm/Group | Electrical Impedance Tomography (EIT) and CO2 Monitor
Number analyzed (Participants) | 8
percentage of total lung space | 71 (11)
Statistical Analysis 1: Comparison: Electrical Impedance Tomography (EIT) and CO2 Monitor; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.09, t-test, 2 sided

9. Secondary Outcome: EIT Metric Functional Lung Space at 32 Weeks Post Menstrual Age in Those Successful in Discontinuation of Non-invasive Ventilation at 33 Weeks Post Menstrual Age.
Description: The first secondary outcome is to determine whether electrical impedance tomography metrics, specifically Global Inhomogeneity Index and Functional Lung Space, measured at 32 weeks post menstrual age are associated with successful discontinuation of non-invasive ventilation at 33 weeks post menstrual age.
Time Frame: as for outcome 3
Population: Data at 32 weeks was available for all 4 infants that weaned to room air at 33 weeks.
Measure: Mean (Standard Deviation); unit: percentage of total lung space
Arm/Group | Electrical Impedance Tomography (EIT) and CO2 Monitor
Number analyzed (Participants) | 4
percentage of total lung space | 79 (8)
Statistical Analysis 1: Comparison: Electrical Impedance Tomography (EIT) and CO2 Monitor; Statistical Analysis assessed correlation of FLS values at 32 weeks between participants that were successful in discontinuation of non-invasive ventilation at 33 weeks postmenstrual age and those that were unsuccessful; Test type: Superiority; p = 0.44, t-test, 2 sided

10. Secondary Outcome: EIT Metric Functional Lung Space at 32 Weeks Post Menstrual Age in Those Unsuccessful in Discontinuation of Non-invasive Ventilation at 33 Weeks Post Menstrual Age.
Description: as for outcome 9
Time Frame: as for outcome 3
Population: Data at 32 weeks was available for 6 of 10 infants that did not wean to room air at 33 weeks
Measure: Mean (Standard Deviation); unit: percentage of total lung space
Arm/Group | Electrical Impedance Tomography (EIT) and CO2 Monitor
Number analyzed (Participants) | 6
percentage of total lung space | 74 (10)
Statistical Analysis 1: Comparison: Electrical Impedance Tomography (EIT) and CO2 Monitor; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.44, t-test, 2 sided

11. Secondary Outcome: EIT Metric Functional Lung Space at 34 Weeks Post Menstrual Age in Those Successful in Discontinuation of Non-invasive Ventilation at 36 Weeks Post Menstrual Age.
Description: The second secondary outcome is to determine whether electrical impedance tomography metrics, specifically Global Inhomogeneity Index and Functional Lung Space, measured at 34 weeks post menstrual age are associated with successful discontinuation of non-invasive ventilation at 36 weeks post menstrual age.
Time Frame: as for outcome 5
Population: Data at 34 weeks was available for 3 of the 4 infants that weaned to room air by 36 weeks
Measure: Mean (Standard Deviation); unit: percentage of total lung space
Arm/Group | Electrical Impedance Tomography (EIT) and CO2 Monitor
Number analyzed (Participants) | 3
percentage of total lung space | 85 (8)
Statistical Analysis 1: Comparison: Electrical Impedance Tomography (EIT) and CO2 Monitor; Statistical Analysis assessed correlation of FLS values at 34 weeks between participants that were successful in discontinuation of non-invasive ventilation by 36 weeks postmenstrual age and those that were unsuccessful; Test type: Superiority; p = 0.59, t-test, 2 sided

12. Secondary Outcome: EIT Metric Functional Lung Space at 34 Weeks Post Menstrual Age in Those Unsuccessful in Discontinuation of Non-invasive Ventilation at 36 Weeks Post Menstrual Age.
Description: as for outcome 11
Time Frame: as for outcome 5
Population: Data at 34 weeks was available for 4 of the 6 infants that did not wean to room air by 36 weeks
Measure: Mean (Standard Deviation); unit: percentage of total lung space
Arm/Group | Electrical Impedance Tomography (EIT) and CO2 Monitor
Number analyzed (Participants) | 4
percentage of total lung space | 81 (8)
Statistical Analysis 1: Comparison: Electrical Impedance Tomography (EIT) and CO2 Monitor; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.59, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from enrollment through study completion which coincides with discharge from NICU at 36-43 weeks postmenstrual age. Depending on birth gestational age and discharge from NICU, adverse events are recorded during a period of 6 weeks (highest eligible birth gestational age to youngest postmenstrual age at NICU discharge) to 18 weeks (lowest possible birth gestational age to oldest postmenstrual age at NICU discharge).
Arm/Group | Electrical Impedance Tomography (EIT) and CO2 Monitor
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
Missing data due to enrollment timing, research staff limitations. The primary outcome is missing data in 9 of 20 infants. The secondary outcomes are missing 4 of 14 and 3 of 10 respectively. There is also potential of measurement error/noise due to variations in belt positioning, infant movement, and interference from respiratory monitoring equipment. The small sample size restricted ability to detect significant differences especially in secondary objectives as few infants analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT06609135/Prot_SAP_004.pdf
  • Informed Consent Form (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/35/NCT06609135/ICF_003.pdf